CLINICAL TRIAL: NCT01013272
Title: Lamivudine Therapy in Patients With Prior Entecavir Treatment and Undetectable Viral Load
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, James Yan Yue Fung, Dr, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HKUHEP-01
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Hepatitis B, Chronic
Keywords: entecavir; lamivudine; sequential therapy
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Entecavir (Active Comparator): Ongoing entecavir 0.5mg daily
  Interventions: Drug: Entecavir
- Lamivudine (Active Comparator): Switch to lamivudine 100mg daily
  Interventions: Drug: Lamivudine

INTERVENTIONS:
Drug: Entecavir — Entecavir 0.5mg orally daily
  Other Names: Baraclude
  Arms: Entecavir
Drug: Lamivudine — Lamivudine 100mg orally, daily
  Other Names: Zeffix
  Arms: Lamivudine

SUMMARY:
Patients with chronic hepatitis B and treated with entecavir for over 6 months (with no previous other antiviral treatment) will be invited to participate in this study. They will be eligible if their liver tests are normal and their viral load is undetectable. Patients will be switched to lamivudine treatment to assess whether lamivudine can maintain adequate suppression of the hepatitis B virus after successful treatment with entecavir. Patients will be monitored closely after switching treatment at 1 months and then every 3 monthly. If there is any evidence of increase in viral load then patients will be given the option of changing back to entecavir.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hepatitis B treated with entecavir for 6 months or more
* Normal ALT
* Undetectable HBV DNA by Roche Taqman PCR Assay
* No other previous therapy with nucleoside/nucleotide analogues

Exclusion Criteria:

* Presence of other liver diseases including hepatitis C co-infection, autoimmune hepatitis , primary biliary cirrhosis, primary sclerosing cholangitis, alcoholic liver disease, and Wilson's disease
* History of hepatocellular carcinoma
* History of decompensated liver disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Determine the efficacy of lamivudine therapy in patients with prior entecavir treatment with undetectable viral load | 96 weeks

SECONDARY OUTCOMES:
Determine the chance of lamivudine resistance in patients with prior entecavir treatment with undetectable viral load | 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James Fung, MBChB, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China